CLINICAL TRIAL: NCT01915602
Title: A Prospective, Single-arm, Multicenter, Uncontrolled, Open-label Phase II Trial of Refametinib (BAY86-9766) in Combination With Sorafenib as First Line Treatment in Patients With RAS Mutant Hepatocellular Carcinoma (HCC)
Brief Title: Refametinib in Combination With Sorafenib in RAS Mutant Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16728; 2013-000241-39 (EudraCT Number)
Record Dates: First submitted 2013-07-24; First posted 2013-08-05 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Carcinoma; Mitogen-activated Extracellular-signal-regulated kinase (MEK) inhibitor; Sorafenib; Objective tumor response rate (ORR); modified RECIST criteria
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — N-(3,4-difluoro-2-(2-fluoro-4-iodophenylamino)-6-methoxyphenyl)-1-(2,3-dihydroxypropyl)cyclopropane-1-sulfonamide; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Refametinib and Sorafenib (Nexavar) (Experimental): In Cycle 1 reduced sorafenib dose (600 mg daily; 200 mg in the morning + 400 mg in the evening) is administered, which is escalated to the standard dose in Cycle 2, if no Hand-foot skin reaction (HFSR), fatigue, or gastrointestinal (GI) toxicities of grade 2 or higher occur. For the purposes of data recording, the treatment period will be divided into 3-week cycles. Patients will continue on treatment until at least one of the following occurs (main criteria): Progressive Disease (PD) {PD as defined by mRECIST criteria or clinical progression [e.g. Eastern Cooperative Oncology Group performance status (ECOG PS) of ≥3], treatment may be continued past radiological progression, provided the patient derives clinical benefit as judged by the treating physician.}, Death, Unacceptable toxicity, Subject withdraws consent, Treating physician determines discontinuation of treatment is in the subject's best interest, Substantial non-compliance with the protocol
  Interventions: Drug: Refametinib (BAY86-9766); Drug: Sorafenib (BAY43-9006)

INTERVENTIONS:
Drug: Refametinib (BAY86-9766) — Patients will receive refametinib 50 mg (2x20 mg + 1x10mg capsules or 50 mg tablets) bid
Drug: Sorafenib (BAY43-9006) — Patients will receive sorafenib 400 mg (2 x 200 mg tablets) bid.

SUMMARY:
This is a study to investigate the potential clinical benefit of refametinib when given in combination with sorafenib as first line treatment in patients with unresectable or metastatic HCC carrying a RAS mutation. The study will be conducted in 2 stages. Approximately 95 patients (15 at Stage 1/ 80 at Stage 2) will be accrued to this study to receive treatment. Stage 2 of the trial will only be conducted if at least 5 out of 15 patients at Stage 1 show at least partial response according to an objective criteria to evaluate tumor size based on contrast enhancement [modified response evaluation criteria in solid tumors (mRECIST)] assessed by external independent radiologists.

Refametenib is an oral (i.e. taken by mouth) protein kinase inhibitor. A kinase inhibitor targets certain key proteins that are essential for the survival of the cancer cell. By specifically targeting these proteins, refametinib in combination with sorafenib may stop cancer growth. The growth of the tumor may be decreased by preventing these specific proteins from functioning.

The primary endpoint (the most meaningful result to be tracked) of this study is based on the rate of response, i.e. the disease getting smaller. The aim is to show that the therapy with refametinib in combination with sorafenib improves the response rate in this patient population compared to historical results observed with the sorafenib only.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for RAS mutation testing

* Unresectable or metastatic HCC, confirmed either by histology or clinically according to the American Association for the Study of Liver Disease (AASLD) criteria for cirrhotic patients. For non-cirrhotic patients, histological confirmation is mandatory.
* Male or female ≥18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance state 0 or 1.
* Life expectancy of at least 12 weeks.
* No prior use of targeted agents, experimental therapy or systemic anti-cancer treatment.
* No previous treatment with sorafenib or refametinib. Criteria for study treatment eligibility
* Patient must harbor GTPase Kirsten rat sarcoma viral oncogene homolog (KRAS) or Neuroblastoma RAS viral oncogene homolog (NRAS) mutation based on Beads, emulsions, amplification, and magnetic technology, sensitive mutation detection (BEAMing) plasma test.
* Patients must have at least one uni-dimensional measurable lesion by Computed tomography (CT) or Magnetic resonance (MR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and Modified Response Evaluation Criteria in Solid Tumors (mRECIST) which is either naïve (not previously treated by local therapy such as surgery, radiation therapy, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation) or previously treated and has progressed until baseline (both measureable lesion and/or progressed lesion have to be confirmed by central image review of baseline and progression scan).
* ECOG performance status of 0 or 1.
* Liver function status of Child-Pugh Class A.
* Adequate bone morrow, liver, and renal function
* Patient has within normal range cardiac function confirmed by the enrolling clinical institute as measured by echocardiogram or multiple gated acquisition (MUGA) scan.
* Patients who are therapeutically anti-coagulated with an agent such as warfarin or heparin are allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists. Close monitoring of at least weekly evaluations will be performed until International normalized ratio (INR) is stable (within Child Pugh class A threshold) based on a measurement at pre-dose, as defined by the local standard of care.

Exclusion Criteria:

* Any Cancer curatively treated < 3 years prior to study entry, except cervical carcinoma in situ (CIS), treated basal cell carcinoma, and superficial bladder tumors [Staging: noninvasive papillary tumor (Ta), CIS carcinoma (Tis) and tumor invades lamina propria (T1)].
* Patients who are eligible for surgery, liver transplantation, ablation or transarterial chemoembolization for HCC.

History of cardiac disease:

* Congestive heart failure New York Heart Association (NYHA) > class 2.
* Unstable angina (angina symptoms at rest, new-onset angina i.e. within the last 3 months) or myocardial infarction (MI) within the past 6 months prior to start of screening.
* Cardiac arrhythmias requiring anti-arrhythmic therapy.
* QTc (corrected QT interval) > 480 ms
* Uncontrolled hypertension (systolic blood pressure [BP] >150 mmHg or diastolic blood pressure >90 mmHg despite optimal medical management).
* Ongoing infection > Grade 2 according to National Cancer Institute - Common Toxicity Criteria for Adverse Events version 4.03 (NCI-CTCAE version 4.03) Hepatitis B is allowed if no active replication (defined as abnormal Alanine aminotransferase [ALT] >2x Upper limit normal [ULN] associated with Hepatitis B virus [HBV] DNA >20,000 IU/mL) is present. Hepatitis C is allowed if no antiviral treatment is required.
* Known history of, or symptomatic metastatic brain or meningeal tumors (head CT or MR at Screening to confirm the absence of central nervous system [CNS] disease if patient had symptoms suggestive or consistent with CNS disease).
* History of interstitial lung disease (ILD).
* History of hepatic encephalopathy.
* History of organ allograft, cornea transplantation will be allowed.
* History or current evidence of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
* Visible retinal pathology as assessed by ophthalmologic exam that is considered a risk factor for RVO or CSR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-09-27 (Actual); Primary Completion 2015-07-29 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Objective tumor response according to Modified Response Evaluation Criteria in Solid Tumors (mRECIST) assessed by central radiological review | Approximately 36 months

SECONDARY OUTCOMES:
Objective tumor response according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by central radiological review | Approximately 36 months
Objective tumor response according to RECIST 1.1 and mRECIST assessed by investigators | Approximately 36 months
Disease control (central and investigator's assessment) | Approximately 36 months
Overall survival | Approximately 36 months
Time to radiographic tumor progression (central and investigator's assessment) | Approximately 36 months
Duration of response (central and investigator's assessment) | Approximately 36 months
Time to objective response (central and investigator's assessment). | Approximately 36 months
Change in tumor size (central and investigator's assessment) | Approximately 36 months
Best overall response (central and investigator's assessment) | Approximately 36 months
Progression-free survival (central and investigator's assessment) | Approximately 36 months
Number of participants with adverse events as a measure of safety and tolerability | Approximately 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (68):
- Louisville, Kentucky, United States
- Vienna, Austria
- Belgium (4):
  - Bruxelles - Brussel
  - Edegem
  - Leuven
  - Liège
- China (3):
  - Guangzhou, Guangdong
  - Beijing
  - Shanghai
- Czechia (2):
  - Hradec Králové
  - Olomouc
- France (8):
  - Bordeaux
  - Caen
  - Lyon
  - Marseille
  - Nice
  - Paris
  - Saint-Priest-en-Jarez
  - Vandœuvre-lès-Nancy
- Germany (7):
  - Heidelberg, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Frankfurt am Main, Hesse
  - Essen, North Rhine-Westphalia
  - Magdeburg, Saxony-Anhalt
  - Berlin
  - Hamburg
- Hong Kong, Hong Kong
- Hungary (4):
  - Budapest
  - Debrecen
  - Pécs
  - Zalaegerszeg
- Israel (4):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
- Italy (3):
  - Bologna, Emilia-Romagna
  - Rome, Lazio
  - Milan, Lombardy
- Japan (10):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Fukuoka, Fukuoka
  - Yokohama, Kanagawa
  - Osakasayama-shi, Osaka
  - Irima-gun, Saitama
  - Bunkyo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Kyoto
  - Osaka
- Auckland, New Zealand
- Singapore, Singapore
- South Korea (3):
  - Seoul, Seoul Teugbyeolsi
  - Daegu
  - Seoul
- Spain (5):
  - Santiago de Compostela, A Coruña
  - L'Hospitalet de Llobregat, Barcelona
  - Vigo, Pontevedra
  - Oviedo, Principality of Asturias
  - Madrid
- Bern, Switzerland
- Taiwan (2):
  - Tainan
  - Taipei
- Thailand (3):
  - Chiang Mai
  - Khon Kaen
  - Songkhla
- Turkey (Türkiye) (2):
  - Istanbul
  - Mersin
- United Kingdom (2):
  - Birmingham
  - London

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/